CLINICAL TRIAL: NCT00576199
Title: A Phase II Single Arm, Multi-centre Study of Bevacizumab (Avastin®) Pre- and Post-transarterial Chemoembolisation (TACE) Treatment for Localized Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Study of Avastin (Bevacizumab) and Transarterial Chemoembolisation (TACE) Treatment in Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21358
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Bevacizumab

ARMS (1):
- Bevacizumab 5 mg/kg (Experimental): Participants received bevacizumab 5 mg/kg intravenously every 2 weeks and within 24-48 hours prior to each transarterial chemoembolization (TACE) until disease progression or unmanageable toxicity. TACE was conducted for 4 sessions at 8-10 week intervals.
  Interventions: Drug: Bevacizumab; Procedure: Transarterial chemoembolisation (TACE)

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a sterile liquid in single-use vials.
  Other Names: Avastin
Procedure: Transarterial chemoembolisation (TACE) — TACE was conducted by the transfemoral artery approach with selective cannulation of the artery supplying the tumor. Cisplatin mixed with Lipiodol in a 1 mg:1 mL ratio was infused intra-arterially up to a maximum dose of 30 mg, depending on tumor size, followed by embolization of the artery using Gelfoam particle until the blood flow slowed. Bilobar lesions were treated by separate catheterization of right and left hepatic arteries followed by injection of the cisplatin-Lipiodol mixture and embolization.
  Patients with stable disease or a partial response after 4 TACE sessions could be given further TACEs upon the investigator's discretion until there was evidence of progressive disease or contraindication due to severe complication or technical failure to perform the TACE.

SUMMARY:
This single-arm, open-label study assessed the efficacy and safety of Avastin (bevacizumab) treatment combined with transarterial chemoembolisation (TACE) in patients with localized unresectable liver cancer. Patients were treated with TACE at 8 or 10 week intervals for 4 sessions (continuation depended on investigator's discretion). Avastin 5 mg/kg intravenously was administered 24-48 hours prior to each TACE session and every 2 weeks between the TACE sessions until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Liver cancer, not suitable for resection.
* At least 1 measurable lesion, and overall tumor lesions occupying < 50% of liver volume
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Patients receiving concurrent radiotherapy or immunotherapy.
* Patients who have received previous chemotherapy, biological agents, or radiotherapy.
* Prior transarterial chemoembolisation (TACE) or transarterial embolisation (TAE).
* Prior liver transplantation or liver resection.
* Current or recent (within 10 days of study start) use of full-dose anticoagulants for therapeutic purposes.
* Patients with high risk esophageal/gastric varices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Hong Kong, Hong Kong

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Participant Flow data are discontinuations from bevacizumab treatment. Data for discontinuations from the study are not available.
Period: Overall Study
Arm/Group | Bevacizumab 5 mg/kg
Started | 30
Completed | 0
Not Completed | 30
Not completed — Adverse Event | 12
Not completed — Insufficient Therapeutic Response | 14
Not completed — Refused Treatment | 2
Not completed — Reason Unspecified | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All participants who received study medication.
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first administration of study drug to the first documented disease progression or death, whichever occurs first. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Months | 11.6 [6.3 to 15.7]

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete response or a partial response. A complete response was defined as the disappearance of all target lesions. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions taking as reference the Baseline sum longest diameter. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. All other lesions (or sites of disease) should be identified as non-target lesions. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Percentage of participants | 23.3 [9.9 to 42.3]

3. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from the first administration of study drug to the first documented disease progression. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. All other lesions (or sites of disease) should be identified as non-target lesions. Target lesions should be selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the longest diameter for all target lesions will be calculated and reported as the Baseline sum longest diameter.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Months | 12.0 [6.3 to 17.1]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first administration of study drug to death.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Months | 19.9 [10.3 to 27.6]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response, Partial Response, or Stable Disease
Description: A complete response was defined as the disappearance of all target lesions. A partial response was defined as at least a 30% decrease in the sum of the LD of target lesions taking as reference the Baseline sum LD. Stable disease was defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions at Baseline. All other lesions (or sites of disease) should be identified as non-target lesions. Target lesions should be selected on the basis of their size (lesions with the LD) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). A sum of the LD for all target lesions will be calculated and reported as the Baseline sum LD.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Percentage of participants | 86.7 [69.3 to 96.2]

6. Secondary Outcome: Tumor Necrosis
Description: Tumor necrosis was quantified in liver lesions greater than 2 cm at Baseline. When MRI showed many cut surfaces for a single tumor, tumor size and the size of necrotic area was measured by accumulation of the serial sections containing the tumor. Lipiodol accumulation in tumor after TACE was regarded as an indication of necrosis. Tumor necrosis was assessed at Baseline and 1 week prior to the next scheduled transarterial chemoembolisation (TACE) for the first 4 TACEs, then 1 week prior to every second TACE till disease progression. The extent of tumor necrosis is presented as the percentage of the tumor volume at Baseline.
Time Frame: Baseline to the end of the study (up to 3 years, 3 months)
Population: Intent-to-treat population: All participants who received study medication.
Measure: Mean (Standard Deviation); unit: Percentage of tumor volume at Baseline
Arm/Group | Bevacizumab 5 mg/kg
Number analyzed (Participants) | 30
Percentage of tumor volume at Baseline
  Lesion 1 (N= 29) | 1.3 (1.00)
  Lesion 2 (N= 11) | 0.8 (0.87)
  Lesion 3 (N= 5) | 1.6 (1.14)
  Lesion 4 (N= 5) | 1.2 (1.30)
  Lesion 5 (N= 4) | 1.0 (1.41)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from enrollment in the study up to 28 days after treatment completion.
Description: Safety population: All participants who received at least 1 dose of study medication.
Arm/Group | Bevacizumab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 17/30
Other Adverse Events (participants affected / at risk) | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 5 mg/kg (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Liver abscess (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Chest discomfort (General disorders) | 2
Pyrexia (General disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hypertension (Vascular disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 5 mg/kg (N=30)
Hypertension (Vascular disorders) | 10
Epistaxis (Vascular disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 2
Injection site haematoma (Injury, poisoning and procedural complications) | 2
Puncture site haemorrhage (Injury, poisoning and procedural complications) | 2
Haemoptysis (Vascular disorders) | 1
Haemorrhoidal haemorrhage (Vascular disorders) | 1
Oesophageal varices (Gastrointestinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Liver abscess (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 2
Wound complication (Injury, poisoning and procedural complications) | 2
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Oesophageal perforation (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Portal vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.